CLINICAL TRIAL: NCT06778785
Title: Game-Based Digital Intervention for Depression in Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pd2402
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Digital Intervention (Smartphone App-based) (Experimental)
  Interventions: Behavioral: Digital Intervention; Other: Personalization Algorithm
- Health Education Placebo (Smartphone App-based) (Placebo Comparator)
  Interventions: Behavioral: Health Education
- Non-personalized Digital Intervention (Smartphone App-based) (Active Comparator)
  Interventions: Behavioral: Digital Intervention

INTERVENTIONS:
Behavioral: Digital Intervention — game-based digital intervention app
  Arms: Non-personalized Digital Intervention (Smartphone App-based); Personalized Digital Intervention (Smartphone App-based)
Behavioral: Health Education — traditional health education app
  Arms: Health Education Placebo (Smartphone App-based)
Other: Personalization Algorithm — a proprietary algorithm that adaptively adjust the treatment module and parameters to personalize the treatment regime
  Arms: Personalized Digital Intervention (Smartphone App-based)

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of digital interventions in treating depression and anxiety in adolescents. The main question it aims to answer is: Can digital interventions effectively alleviate symptoms of depression and anxiety in adolescents? The trial will include a comparison group where researchers will compare the effects of the digital intervention to traditional health education methods to assess their relative efficacy.

Participants will be asked to engage with the digital intervention platform for a period of two months.

ELIGIBILITY:
Inclusion Criteria:

* The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) will be used to assess participants' eligibility based on the diagnostic criteria for depression outlined in the DSM-5(the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition).
* no prior use of antidepressants or antipsychotic medications.
* having a HAMD (Hamilton Depression scale) score >= 8 upon enrollment
* demonstrate normal cognitive function.
* voluntarily agree to participate in the study, and both they and their legal guardians must provide informed consent.
* being able to read and typeset Chinese.

Exclusion Criteria:

* with severe consciousness disorders and a history of psychiatric illness, traumatic brain injury, substance dependence, or acute poisoning
* with concurrent psychiatric disorders (as determined by clinical assessment)
* at high risk of suicide

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 450 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Depression on the 50-point 16-item Hamilton Depression Rating Scale (HAM-D) at Week 8 | baseline and immediately after 8-week intervention
  HAM-D is a clinician-administered depression assessment scale. To adapt to adolescent participants, item 14 (genital symptoms) was removed. Thus, the score was calculated based on the 16 items. Possible scores range from 0 (no symptoms) to 50 (worst symptom). Change = (Week 8 Score - Baseline Score).
Response Rate - 50 Percent or Greater Reduction in the 50-point 16-item Hamilton Depression Rating Scale (HAM-D) at Week 8 | baseline and immediately after 8-week intervention
  HAM-D is a clinician-administered depression assessment scale. To adapt to adolescent participants, item 14 (genital symptoms) was removed. Thus, the score was calculated based on the 16 items. Possible scores range from 0 (no symptoms) to 50 (worst symptom). The response rate was defined as the number of participants with a 50% or greater reduction in HAM-D score from baseline to week 8.

SECONDARY OUTCOMES:
Change from Baseline in ADHD on the 54-point 18-item ADHD Rating Scale-IV | baseline and immediately after 8-week intervention
  ADHD RS IV is a clinician-administered ADHD assessment scale. Possible scores range from 0 (no symptoms) to 50 (worst symptom). Change = (Week 8 Score - Baseline Score).
Change from Baseline in the 7-point Clinical Global Impressions-Severity Scale (CGI-S) | baseline and immediately after 8-week intervention
  CGI-S is a clinician-administered symptom severity scale. Possible scores range from 1 (least severe) to 7 (most severe). Change = (Week 8 Score - Baseline Score).
Change from Baseline in the 88-point 22-item Ruminative Responses Scale (RRS) | baseline and immediately after 8-week intervention
  Rumination is the process of compulsively focused attention on the symptoms of one's distress, and on its possible causes and consequences, as opposed to its solutions. RRS is a self-report scale that measures rumination. Possible scores range from 22 (least ruminative symptoms) to 88 (worst ruminative symptoms). Change = (Week 8 Score - Baseline Score).
Change from Baseline in the 35-point 5-item Satisfaction with Life Scale (SWLS) | baseline and immediately after 8-week intervention
  The SWLS is a short 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. Possible scores range from 5 (lowest satisfaction) to 35 (highest satisfaction). Change = (Week 8 Score - Baseline Score).
The 7-point Clinical Global Impressions-Improvement Scale (CGI-I) | immediately after 8-week intervention
  CGI-S is a clinician-administered total improvement scale. Possible scores range from 1 (very much improved) to 7 (Very much worse).
Change from Baseline in Anxiety on the 52-point 13-item Hamilton Anxiety Rating Scale (HAM-A) at Week 8 | baseline and immediately after 8-week intervention
  HAM-A is a clinician-administered anxiety assessment scale. To adapt to adolescent participants, item 12 (genitourinary symptoms) was removed. Thus, the score was calculated based on the 13 items. Possible scores range from 0 (no symptoms) to 52 (worst symptom). Change = (Week 8 Score - Baseline Score).
Response Rate - 50 Percent or Greater Reduction in the 52-point 13-item Hamilton Anxiety Rating Scale (HAM-A) at Week 8 | baseline and immediately after 8-week intervention
  HAM-A is a clinician-administered anxiety assessment scale. To adapt to adolescent participants, item 12 (genitourinary symptoms) was removed. Thus, the score was calculated based on the 13 items. Possible scores range from 0 (no symptoms) to 52 (worst symptom). Change = (Week 8 Score - Baseline Score). The response rate was defined as the number of participants with a 50% or greater reduction in HAM-D score from baseline to week 8.

OTHER OUTCOMES:
Change from Baseline in Chinese Exam Score at Week 8. | baseline and immediately after 8-week intervention
  The Chinese exam score was obtained by asking the participants the score (standardized to a 100-point scale) of their most recent exam on the subject of Chinese taken at school. Possible scores range from 0 (worst academic performance) to 100 (best academic performance). Change = (Week 8 Score - Baseline Score).
Change from Baseline in Math Exam Score at Week 8. | baseline and immediately after 8-week intervention
  The Math exam score was obtained by asking the participants the score (standardized to a 100-point scale) of their most recent exam on the subject of Math taken at school. Possible scores range from 0 (worst academic performance) to 100 (best academic performance). Change = (Week 8 Score - Baseline Score).
Change from Baseline in English Exam Score at Week 8. | baseline and immediately after 8-week intervention
  The English exam score was obtained by asking the participants the score (standardized to a 100-point scale) of their most recent exam on the subject of English taken at school. Possible scores range from 0 (worst academic performance) to 100 (best academic performance). Change = (Week 8 Score - Baseline Score).

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuang, China